CLINICAL TRIAL: NCT03249259
Title: The Effect of Choline Alfoscerate on Improvement of Cognitive Function in Elderly Patients With Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1508-312-006
Record Dates: First submitted 2017-08-09; First posted 2017-08-15 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glycerylphosphorylcholine; Choline

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind placebo controlled study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choline alfoscerate (Experimental): choline alfoscerate 400mg (2 caps - 1 cap bid)
  Interventions: Drug: Choline alfoscerate
- Control (Placebo Comparator): Placebo (2 caps - 1 cap bid)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Choline alfoscerate — Treatment duration is 6 months and can be extended to 12 months with participant's agreement.
  Other Names: Choline
  Arms: Choline alfoscerate
Drug: Placebo — Treatment duration is 6 months and can be extended to 12 months with participant's agreement.
  Arms: Control

SUMMARY:
In this study, the investigators are going to investigate the efficacy of choline alfoscerate on improvement of cognitive function assessed by MMSE compared to plaebo.

DETAILED DESCRIPTION:
The investigators will enroll patients with type 2 diabetes whose age is equal to higher than 60, and randomly assigned study drug or placebo at 1:1 ratio. The treatment duration is 6 months and extension study will be continued to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* baseline MMSE score 25-28

Exclusion Criteria:

* type 1 diabetes
* diabetes ketoacidosis or hyperosmolar hyperglycemic crisis
* HbA1c over than 9.0%
* MMSE less than 25
* abnormal TSH levels
* vitamin B12 deficiency
* severe infection, perioperative state, trauma
* hypopituitarism or adrenal insufficiency
* any conditions that lead to hospitalization
* chronic alcoholics within 1 year
* any drugs that can influence to cognitive function within 3 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 6 months
  Change of MMSE Score

SECONDARY OUTCOMES:
Glucose metabolism | 6 months
  Changes in HbA1c
Glucose metabolism | 6 months
  Changes in fasting glucose concentration

OTHER OUTCOMES:
Hypoglycemia | 6 months
  Incidence of hypoglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No